CLINICAL TRIAL: NCT03465813
Title: Reducing Distress and Depressive-symptoms in Rural Women Using CaringGuidance™-After Breast Cancer Diagnosis: Randomized Controlled Pilot Study
Brief Title: Reducing Distress and Depressive-symptoms in Rural Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0140-17-EP
Record Dates: First submitted 2018-02-28; First posted 2018-03-14 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer; Psychological Adjustment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CaringGuidance Intervention (Experimental): Three months of web-based CaringGuidance psychoeducational program use, independently on home computer in addition to usual care.
  Interventions: Behavioral: CaringGuidance After Breast Cancer Diagnosis
- Usual Care (No Intervention): Three months of care as usual from subjects' clinics and community as the subject chooses.

INTERVENTIONS:
Behavioral: CaringGuidance After Breast Cancer Diagnosis — CaringGuidance After Breast Cancer Diagnosis, psychoeducational, Internet-accessible program
  Arms: CaringGuidance Intervention

SUMMARY:
Approximately 30% of U.S. breast cancer survivors experience significant cancer-related distress ranging from adjustment disorders, depression-symptoms and major depression up to 20 years after diagnosis. For rural cancer survivors, lack of access to care, support and stigma associated with cancer and mental health, challenge rural women's ability to prevent cancer-related distress and its deleterious outcomes. However, these barriers may be overcome by a new Internet-based psychoeducational program designed for newly diagnosed women; CaringGuidance™- After Breast Cancer Diagnosis. This self-guided program provides information, cognitive-behavioral and supportive coping strategies in a text/audio/visual format accessed via Internet/mobile devices to increase understanding and provide supportive tools to prevent/manage distress and depressive-symptoms. This pilot study will determine preliminary efficacy of the CaringGuidance™ program on distress and depressive-symptoms monthly and over 3 months, for rural women newly diagnosed with breast cancer.

DETAILED DESCRIPTION:
Of the 3.1 million U.S. breast cancer survivors, approximately 30% experience significant cancer-related distress ranging from sub-threshold to diagnosable adjustment disorders, depression-symptoms and major depression up to 20 years after diagnosis. Rural cancer survivors report poorer mental health than urban survivors. Lack of access to care, support and stigma associated with cancer and mental health, challenge rural women's ability to prevent cancer-related distress and its deleterious outcomes. These barriers may be overcome by a new Internet-based, psychoeducational program designed for newly diagnosed women; CaringGuidance™- After Breast Cancer Diagnosis. This self-guided program provides information, cognitive-behavioral and supportive coping strategies in a text/audio/visual format accessed via Internet/mobile devices to increase understanding, and provide supportive tools to prevent/manage distress and depressive-symptoms.

The aims of this pilot study are to determine preliminary efficacy of the CaringGuidance™ program on distress and depressive-symptoms monthly and over 3 months, for rural women newly diagnosed with breast cancer, and trial measures and methods, prior to a fully powered randomized controlled clinical trial.

Sixty rural women, will be randomized to 3 months of self-guided CaringGuidance™ program access with usual care or usual care alone. Both groups complete monthly standard psychosocial measures, daily activity/symptom logs and receive a monthly call. Program engagement/dose will be measured by the CaringGuidance™ internal data system. Descriptive and inferential statistics will characterize the sample and determine differences between groups at monthly intervals and overall. Variability of outcome variables will also be assessed to determine usefulness.

ELIGIBILITY:
Inclusion Criteria:

* experiencing their first, stage 0 - IIIA breast cancer diagnosis (either clinical or definitive early stage at enrollment), and be 19 to 85 years of age,
* enroll < 3 months post-diagnosis (as soon as possible after diagnosis is desirable),
* reside in a non-metro county of the United States according to the USDA Rural-Urban Continuum Codes (6 -9) (RUCC) or at a rural zip-code by the USDA Rural Urban Commuting Area (RUCA) codes (4.0, 4.2, 5.0, 5.2, 6.0, 6.1, 7.0, 7.2-4, 8.0, 8.2-4, 9.0-2, 10.0, 10.2-6)
* be able to read and write in English since the CaringGuidance™ program is in English,
* have regular access (e.g. home or work) to high speed/satellite broadband Internet on desk/laptop or wireless iPad, Android or iPhone throughout the 3 months of the study,*
* have an email address at which to receive CaringGuidance™ prompts,
* have a Baseline Distress Thermometer score of > 4, or an Impact of Events Scale score of > 9, or Center for Epidemiological Studies Depression Scale score of > 16 (i.e. clinically meaningful thresholds).
* Able to comprehend and provide informed consent

Exclusion Criteria:

* Men and women with recurrent or advanced breast cancer
* Those mentally or physically unable to read the consent form or other study materials and/or participate in the consent and engagement with the CaringGuidance program. Women who have been hospitalized for mental health issues or substance abuse in the past year are ineligible.

Ages: 19 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2019-05-11 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
change from baseline in distress at 1, 2, and 3 months | at baseline and months 1, 2, and 3
  self-report of psychological distress
change from baseline in depressive-symptoms at 1, 2, and 3 months | at baseline and months 1, 2, and 3
  self-report of depressive-symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Robin M Lally, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Oncology Clinics, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No